CLINICAL TRIAL: NCT02734979
Title: Prospective Evaluation of a Surgical Solution for Breast Cancer-Associated Lymphedema
Acronym: Biobridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-37161; BRS0095 (Other: OnCore)
Record Dates: First submitted 2016-04-05; First posted 2016-04-12 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Lymphedema; Edema
Keywords: lymphedema; edema
MeSH Terms: conditions — Lymphedema; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Biobridge and lymph node transfer (Experimental): The investigators will investigate whether addition of the Biobridge scaffold to the standard surgery for vascularized lymph node transfer will improve the outcome of surgical treatment in lymphedema of the upper arm. The investigators will perform lymph scans (lymphoscintigrams) before surgery and one year following surgery to determine the success of the surgery. In addition, the volume of the operated arm will be monitored by repeated measurement with a tape measure. The investigators will also track bioimpedance, a painless technique to detect fluid in the tissues. The investigators will obtain small skin biopsies and blood samples to detect the biological changes that may occur as a result of successful surgery.
  Interventions: Device: Biobridge and lymph node transfer

INTERVENTIONS:
Device: Biobridge and lymph node transfer — Biobridge is surgically implanted with conventional vascularized lymph node transfer surgery

SUMMARY:
To investigate whether addition of the Biobridge scaffold to the standard surgery for vascularized lymph node transfer will improve the outcome of surgical treatment in lymphedema of the upper arm.

DETAILED DESCRIPTION:
The investigators will perform lymph scans (lymphoscintigrams) before surgery and one year following surgery to determine the success of the surgery. In addition, the volume of the operated arm will be monitored by repeated measurement with a tape measure. The investigators will also track bioimpedance, a painless technique to detect fluid in the tissues. The investigators will obtain small skin biopsies and blood samples to detect the biological changes that may occur as a result of successful surgery.

ELIGIBILITY:
Inclusion Criteria:

The subject must be a breast cancer survivor, at least three years beyond completion of cancer therapy, free of clinical disease, and eligible for surgical intervention.

* Ages 18 to 75 years (inclusive).
* Swelling of 1 limb that is not completely reversed by elevation or compression
* Stage II or greater lymphedema at screening, based on the International Society of Lymphology (ISL) staging system
* Completion of a full course of complete decongestive therapy (CDT), according to ISL guidelines at least 8 weeks prior to screening, including use of compression garments for at least 8 weeks without change in regimen
* Willingness to maintain a stable regimen of self-care, with consistent use of compression garments from screening through the entire study duration (through the safety follow-up visit). Self-bandaging, use of nighttime compression garments, and intermittent pneumatic compression devices are allowed, but the procedures and regimens must remain consistent from screening though the entire study duration.
* Two consecutive measurements of limb volume (LV) in the affected limb taken at least 1 day apart during the screening period must be within 10% of each other. A maximum of 3 measurements can be taken. Affected limb volume ratio >20% (affected limb compared to unaffected limb); volume measurements will be performed and volume ratio will be calculated at S1 and S2 visit.
* Evidence of abnormal bioimpedance ratio, if feasible based upon unilateral disease: L-Dex >10 units; bioimpedance performed at S1 and S1
* Willingness and ability to understand and the willingness to sign a written informed consent form document
* Willingness and ability to comply with all study procedures, including measurement of skin thickness using skin calipers.
* Participants must have NED, completed breast cancer therapy 3 years prior to enrollment.
* ECOG 0- 2

Exclusion Criteria:

* Edema arising from increased capillary filtration will be excluded.
* Inability to safely undergo general anesthesia and/or perioperative care related to vascularized lymph node transfer
* Concurrent participation in a clinical trial of any other investigational drug or therapy, regardless of indication, within 1 month before screening or 5 times the drug's half-life, whichever is longer
* Recent initiation of (≤8 weeks), or intention to initiate, CDPT or maintenance physiotherapy for lymphedema at any time during the duration of the study
* Other medical condition that could lead to acute limb edema, such as (but not limited to) acute venous thrombosis
* Other medical condition that could result in symptoms overlapping those of lymphedema in the affected limb (e.g., pain, swelling, decreased range of motion)
* History of clotting disorder (hypercoagulable state)
* Chronic (persistent) infection in the affected limb
* Any other infection (unrelated to lymphedema) within 1 month prior to screening
* Current evidence of malignancy or any high risk for breast cancer recurrence (Stage III or IV, ER/PR/HER-2 negative (triple negative) cancer , locally advanced disease, inflammatory breast cancer, > 3 positive axillary lymph nodes, extracapsular nodal extension, invasive micropapillary breast carcinoma, or if performed, patients with a high risk of recurrence based on multi-gene signatures, e.g. BRCA1, BRCA 2, Oncotype DX (high risk recurrence score) or Mammaprint (poor risk signature)
* Currently receiving chemotherapy or radiation therapy
* Life expectancy < 2 years for any reason
* Pregnancy or nursing
* Substance abuse (such as alcohol or drug abuse) within 6 months prior to screening
* Significant or chronic renal insufficiency (defined as serum creatinine > 2.5 mg/dL or an estimated glomerular filtration rate [eGFR] < 30 mL/min at screening) or requires dialytic support
* Hepatic dysfunction, defined as alanine transaminase (ALT) or aspartate transaminase (AST) levels > 3 × upper limit of the normal range (ULN) and/or bilirubin level > 2 × ULN at screening
* Absolute neutrophil count < 1500 mm3 at screening
* Hemoglobin concentration < 9 g/dL at screening
* Known sensitivity to porcine products
* Any reason (in addition to those listed above) that, in the opinion of the investigator, precludes full participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biobridge and Lymph Node Transfer
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biobridge and Lymph Node Transfer
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Limb Volume
Description: Lymphoscintigraphy, a measure of limb volume indicative of adequate limb drainage, was conducted on the arm receiving BioBridge implantation (affected arm) and the contralateral (unaffected) arm, before surgery (baseline) and 1 year following surgical implantation of the Biobridge device. The outcome is reported as the median difference in the pre-implantation baseline value and the value 1 year after surgery for each arm.
Time Frame: 1 year
Population: The units analyses are the affected arm (received BioBridge implant) and the unaffected contralateral arm.
Measure: Number; unit: mL
Arm/Group | Biobridge and Lymph Node Transfer
Number analyzed (Participants) | 1
mL
  BioBridge implant arm | -15
  Unaffected contralateral arm | -202

2. Secondary Outcome: Serial Lymphoscintigraphy (LSG)
Description: Lymphoscintigraphy, a measure of limb volume for which changes are indicative of adequate limb drainage, was conducted on the arm receiving the BioBridge implantation (baseline) and 1 year following the Biobridge implantation. The outcome is reported as the median difference in measured volume for affected arm from baseline to 1 year.
Time Frame: 1 year
Measure: Number; unit: mL
Arm/Group | Biobridge and Lymph Node Transfer
Number analyzed (Participants) | 1
mL
  Baseline | 2295
  1 year | 2280

3. Secondary Outcome: Bioimpedance Spectroscopy
Description: Bioimpedance spectroscopy (BIS) is a non-invasive technique to measure the volume of fluid in various parts of the body, and can be used to assess the extent of lymphedema. BIS involves passing an extremely low-strength electrical current through the area and measuring how the flow of the current is slowed by the fluid in the body, and is reported as Ri in ohms, meaning the resistance of the intracellular fluid. BIS was conducted on the arm with the BioBridge implant, at baseline and 1 year after surgery. The outcome is reported as the median difference between baseline and 1 year after surgery in the arm receiving the BioBridge implant.
Time Frame: 1 year
Measure: Number; unit: ohms
Arm/Group | Biobridge and Lymph Node Transfer
Number analyzed (Participants) | 1
ohms
  Baseline | 951.8
  1 year | 977.3

4. Secondary Outcome: Caliper Skin-fold Thickness
Description: Skin fold thickness as measured by calipers was used as a measure of fluid retention. Skin fold thickness was measured at the upper arm, forearm, and back of the hand, at baseline and at 1 year following surgical implantation of the Biobridge device. An increase in skin thickness means increased fluid retention. The outcome is reported as the median difference of skin fold thickness in millimeters (mm) for each location on the arm receiving the BioBridge implant, from baseline to 1 year.
Time Frame: 1 year
Measure: Number; unit: millimeters (mm)
Units Other Than Participants: Skin-fold location
Groups:
- Caliper Skin-fold Thickness - Upper Arm: Caliper skin-fold thickness as measured at the upper arm, of the arm receiving the BioBridge implant.
- Caliper Skin-fold Thickness - Forearm: Caliper skin-fold thickness as measured at the forearm, of the arm receiving the BioBridge implant.
- Caliper Skin-fold Thickness - Hand: Caliper skin-fold thickness as measured on the back of the hand, of the arm receiving the BioBridge implant.
Arm/Group | Caliper Skin-fold Thickness - Upper Arm | Caliper Skin-fold Thickness - Forearm | Caliper Skin-fold Thickness - Hand
Number analyzed (Participants) | 1 | 1 | 1
Number analyzed (Skin-fold location) | 1 | 1 | 1
millimeters (mm)
  Baseline | 2.5 | 3.5 | 2.5
  1 Year | 3.25 | 3.25 | 2.25

5. Secondary Outcome: Cutaneous Punch Biopsy of Skin
Description: Serial changes in histopathology will be determined via a blinded assessment of serial cutaneous punch biopsies specimens.
Time Frame: 1 year
Population: The per-protocol analysis was specified to be a blinded analysis, but with only a single set of specimens the analysis could not be conducted as defined.
Arm/Group | Biobridge and Lymph Node Transfer
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life for Limb Lymphoedema (LYMQOL)
Description: Quality-of-life was assessed using the LYMQOL survey, a 5-question survey for improved function, appearance, symptoms, mood, and overall QOL. Overall QoL was reported on a 10-point scale with 10 being best, and the other assessments were for disease impact on a 4-point response scale consisting of 1 (none), 2 (a little), 3 (quite a bit), 4 (a lot), with lower values representing minimal disease (lymphedema) impact on the parameter and higher values representing a greater negative effect on the parameter. The outcome is reported as the median.
Time Frame: 1 year
Measure: Number; unit: units on a scale
Groups:
- LYMQOL Survey - Overall QoL: LYMQOL Survey for overall quality of life (QoL) after receiving the BioBridge implant. Survey is a 10-point scale.
- LYMQOL Survey - Function: LYMQOL Survey for function in the arm receiving the BioBridge implant. Survey is a 4-point scale.
- LYMQOL Survey - Appearance: LYMQOL survey for appearance of the arm receiving the BioBridge implant. Survey is a 4-point scale.
- LYMQOL Survey - Symptoms: LYMQOL survey for lymphedema symptoms in the arm receiving the BioBridge implant. Survey is a 4-point scale.
- LYMQOL Survey - Mood: LYMQOL survey for mood after receiving the BioBridge implant. Survey is a 4-point scale.
Arm/Group | LYMQOL Survey - Overall QoL | LYMQOL Survey - Function | LYMQOL Survey - Appearance | LYMQOL Survey - Symptoms | LYMQOL Survey - Mood
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
units on a scale
  Baseline | 7 | 2.2 | 3.4 | 2.6 | 1.4
  1 year | 9 | 1.2 | 1.6 | 1.5 | 1.3

ADVERSE EVENTS:
Time Frame: 2 years 8 months
Arm/Group | Biobridge and Lymph Node Transfer
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biobridge and Lymph Node Transfer (N=1)
Edema (Cardiac disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT02734979/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT02734979/ICF_001.pdf